CLINICAL TRIAL: NCT02721134
Title: Diagnostic Performance of a New Bio-marker During Bacterial Sepsis
Acronym: BACTIDIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Bio-Rad Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-PP-18
Record Dates: First submitted 2016-03-07; First posted 2016-03-29 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- additional blood tubes (Other)
  Interventions: Other: additional blood tubes

INTERVENTIONS:
Other: additional blood tubes — four whole blood tubes 5 ml (2 + EDTA tubes separating gel and dry tubes 2 + separating gel ) will be taken in order to assay more bacterial biomarkers on day 0 , J1, J2, J3 and J5

SUMMARY:
Sepsis is a constant concern in ICU, frequent and severe, it requires early diagnosis and prompt implementation of the etiological treatment. The bacterial infections are the most common and are associated with high morbidity and mortality. Diagnosis is based on the detection of micro-organisms (bacteria) that can confirm the diagnosis and to tailor antibiotic treatments. Blood cultures are positive in 30-35% of cases and diagnosis is often based on a body of evidence that the use of biomarkers. No biomarkers (or even a combination of biomarkers) no evidence to confirm or refute the diagnosis of sepsis alone. During sepsis, gram + and gram - are circulating and often present in small amounts; they can be detected by sensitive and specific tools following a pretreatment of the blood sample (innovative technology Bacti-DIAG).

The main objective of the multicentre study Bacti-DIAG-Rea is testing in prospectively, in a suspicious population resuscitation of sepsis, this new bacterial biomarker. Secondary objectives will assess whether Bacti-DIAG provides time and precision gain (gram + vs grams) in the patient's care including diagnosis and treatment.

All ICU patients and with clinical criteria of Systemic Inflammatory Response Syndrome (SIRS) sepsis suspects will be included: in addition to the samples taken for routine care of the patient 4 tubes of whole blood will be collected 5mL. The definitive diagnosis of sepsis or SIRS be confirmed retrospectively by two independent experts blinded to Bacti-DIAG. The areas under the ROC curves for the detection of gram + and gram will be calculated and associated detection limits will be determined to meet the objectives of the study.

It is planned to include 400 consecutive patients with SIRS criteria for sepsis 300-360 and analyze biometric and biological data based on the subsequent evolution of the patients. The care of patients will be blinded to the results of the new biomarker Bacti-DIAG

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years
* Patient hospitalized in ICU with a diagnosis of SIRS:
* Temperatures above 38 ° C or below 36 ° C

At least one other criterion from:

* Heart rate> 90 bpm
* Respiratory rate above 20 breaths / min or PaCO2 <32 mmHg
* Leukocytosis greater than or less than 4000/mm3 12000/m3

  * Patient admitted in intensive care for less than 12 hours
  * Patient does not preclude its participation in the study.

Exclusion Criteria:

* No affiliation to a social security scheme (beneficiary or assignee)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
determine the AUC | 2 years
  determine the AUC of a test ( Bacti DIAG ) for the diagnosis of sepsis and sepsis Gram + Gram - relative to the composite gold standard . Two analyzes will be performed , one for the diagnosis of sepsis Gram + and to that of sepsis Gram . We describe below the analysis to be conducted on Gram + diagnosis , it will suffice to transpose the study of Gram

CONTACTS AND LOCATIONS:
Locations (6):
- France (5):
  - Antibes hospital Center, Antibes
  - Cannes Hospital, Cannes
  - Draguignan Hospital, Draguignan
  - Frejus Hospital, Fréjus
  - CHU de Nice, Nice
- Monaco princesse grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No